CLINICAL TRIAL: NCT03163719
Title: Impact of Early Lactate Dosage Compared to CK for Diagnosis of a Suspected Seizure, on Patient Admitted to an Emergency Unit
Brief Title: Impact of Early Lactate Dosage Compared to CK for Diagnosis of a Suspected Seizure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-329
Record Dates: First submitted 2017-05-09; First posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Epileptic Seizure; Creatine Kinase; Lactate; Epileptic Generalized Tonic-clonic Seizure
Keywords: Seizure; Generalized convulsive seizure; Convulsions; Creatine Kinase; Lactate; Lactacidaemia; Diagnostic; Losing consciousness; Epilepsy; Epileptic generalized tonic-clonic seizure
MeSH Terms: conditions — Seizures; Epilepsy, Generalized; Disease; Epilepsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with generalized convulsive seizure: All adult patients (aged at least 18 years old) presenting to the CHU Clermont-Ferrand adult emergencies with a strong suspicion of generalized tonic-clonic seizure beginning less than 4 hours will be included. Each eligible patient will be proposed by a doctor, to participate to the study. The emergency doctor will verify the patient's inclusion and non-inclusion criteria.
  Interventions: Diagnostic Test: CK and Lactate dosages

INTERVENTIONS:
Diagnostic Test: CK and Lactate dosages — A patient consulting the emergency department for suspected seizure will have an usual blood test at the admission in this context with notably ionogram, fasting glucose, venous gasometry. As the CHU purchased a venous and arterial gasometry reader for the emergency department, blood ionogram, Hb, lactates, HCO3-, pH are collected without delay. The Creatine kinase dosage will be collected in the usual way as a "tube bottom". As recommended by the French Society of Neurology, a new sample will be collected at 4 hours of seizure for a dosage of Creatine kinase. The determination of the lactates will be based on a "tube bottom".

SUMMARY:
Defining the origin of a seizure remains a difficult diagnosis. The presence of witness is not systematic, the clinical examination can be little contributory, and the delay recommended by the FSN is often surpassed for the realization of Creatine kinase (4h). In the event of a suspected seizure, an initial blood test with Creatine kinase and Lactates is often done on admission of the patient in other words before the 4hours delay.

It seems interesting to harmonize the practices, to limit the patient wait in the emergencies for a deferred dosage of CK at 4 hours from the seizure and to identify an early biological marker.

Objectives:

To evaluate the value of blood CK and Lactate dosage in emergency procedures in the diagnosis of generalized seizures.

DETAILED DESCRIPTION:
We propose to carry out a prospective, observational, monocentric study at the CHU of Clermont-Ferrand. This is a descriptive analysis of the kinetics of the Creatine kinase and Lactates rates collected at the admission of a patient consulting for strong suspicion of convulsive seizure, and at 4 hours from the generalized seizure.

A patient consulting the emergency department for suspected seizure will have an usual blood test at the admission in this context with notably ionogram, fasting glucose, venous gasometry. As the CHU purchased a venous and arterial gasometry reader for the emergency department, blood ionogram, Hb, lactates, HCO3-, pH are collected without delay.

The Creatine kinase dosage will be collected in the usual way as a "tube bottom".

As recommended by the French Society of Neurology, a new sample will be collected at 4 hours of seizure for a dosage of Creatine kinase. The determination of the lactates will be based on a "tube bottom".

It is the emergency practitioner who will decide whether or not to include the patient in the descriptive study, assisted by a standardized survey, enumerating the high probability of generalized seizure orientation characteristics (patient history, treatments including antiepileptics, anamnesis, witnesses presence, evocative clinic) The study only recruited cases of strong suspicion of generalized seizure, beginning less than 4 hours to compare the kinetics of Creatine kinase and Lactates at admission and 4 hours of the generalized seizure.

ELIGIBILITY:
Inclusion Criteria:

* Any generalized convulsive seizure defined by a transient loss of consciousness with the occurrence of tonic-clonic movements.
* Beginning less than 4 hours.
* In a highly evocative context of the crisis by the presence of: witnesses and/or Urine loss, Tongue bite and/or personal medical history of epilepsy and/or Favorable context: sleeping debt, drug withdrawal, lights stimulations, video games and/or Impression of "already lived", already experienced before the discomfort and/or Break contact, and/or Unusual posture with hypertonia and/or Amnesia of the episode and/or Post-episode Confusion
* Inaugural or recurrent

Exclusion Criteria:

* Patient Refusal
* <18 years
* Pregnancy
* Sepsis, fever> 38 °
* Shock State
* Myocardial infarction
* Unbalanced Diabetes
* Hepatocellular insufficiency
* Drug and Toxic Use
* Taking Metformin
* Significant muscle injuries
* Myopathy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients (aged at least 18 years old) presenting to the CHU Clermont-Ferrand adult emergencies with a strong suspicion of generalized tonic-clonic seizure beginning less than 4 hours will be included. Each eligible patient will be proposed by a doctor, to participate to the study. The emergency doctor will verify the patient's inclusion and non-inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-11-28 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Comparison of lactates measurement and CPK measurement | Less than 4 hours
  at admission and four hour after admission for a confirmed convulsive crisis

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, Auvergne, France